CLINICAL TRIAL: NCT06091839
Title: Anchor Versus Parachute Suturing Technique in Arteriovenous Fistula Creation for Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Abdullah Yahya Mohamed Fouda, Vascular surgery specialist, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MKSU 50-12-8
Record Dates: First submitted 2023-10-11; First posted 2023-10-19 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Arterio-venous Fistula
MeSH Terms: conditions — Arteriovenous Fistula | interventions — Suture Techniques; Renal Dialysis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- anchor technique (Active Comparator): In the anchor technique , the suture was secured first at the heel region after entering the artery and the vein in an inside-out fashion, and a surgical knot was tied, after which the suture was run continuously across the lateral margins of anastomosis, entering the vein outside-in and the artery inside-out, from heel (proximal end of arteriotomy) to toe (distal end). Then the suture was run to complete suturing the medial margins from heel to toe, entering the artery outside-in and the vein inside-out, and final knots were taken.
  Interventions: Other: suturing technique in arteriovenous fistula creation for hemodialysis
- parachute technique (Active Comparator): In the parachute technique, suture was first secured at 11 o'clock position entering both vessels in an inside-out fashion, then continuous suturing was commenced towards 5 o'clock position across the heel, entering the vein outside-in and the artery inside-out, without approximating the vessels. Then, gentle traction was applied on the sutures to allow even distribution of tension along the suture-line and 'parachuting' or approximation of vessel walls together. The suture was then run in a continuous fashion across the proximal margin (toward surgeon) and across the toe region, and finally, surgical knots were applied at midway on the distal margin.
  Interventions: Other: suturing technique in arteriovenous fistula creation for hemodialysis

INTERVENTIONS:
Other: suturing technique in arteriovenous fistula creation for hemodialysis — End-to-side AV anastomosis was created in upper limb between cephalic vein and brachial or radial artery

SUMMARY:
Randomized controlled study to compare the results of two surgical techniques for AVF creation, including the anchor technique (Group A) and parachute technique (Group B).

The study population will be patients referred to the Vascular surgery department for the creation of Hemodialysis access. Patients will be advised to undergo elective surgery for AVF once their renal Glomerular Filtration Rate Estimated (eGFR) is less than 15 ml/min.

primary outcome: Functional Maturation of Arterio-venous Fistula [ Time Frame: Six Months] Ready fistula for cannulation, vein length at least 10 cm, diameter more than 6 mm, depth not more than 6 mm, and ability of the access to deliver a flow rate of 600ml/min and maintain dialysis for 4 hours.

DETAILED DESCRIPTION:
Introduction

Aim of the work To compare the results of two surgical techniques for AVF creation, including the anchor technique (Group A) and parachute technique (Group B).

Patients and the method Study location: We will submit the study protocol for approval by Kafr ElSheikh medical research ethics committee, faculty of medicine, Kafr ElSheikh University.

Study design: Randomized controlled study will be conducted in the department of vascular surgery in Kafr El Sheikh.

Time of study: We started in march 2022.

Study population: The study population will be patients referred to the Vascular surgery department for the creation of Hemodialysis access. Patients will be advised to undergo elective surgery for AVF once their renal Glomerular Filtration Rate Estimated (eGFR) is less than 15 ml/min.

The number of patients:

This study will be done on 150 cases, 75 cases in group A (anchor technique) and another 75 in group B (parachute technique).

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years of age or older.
* Need for AVF creation for vascular access for planned hemodialysis (within one year), Including distal - Radio-cephalic, proximal brachio-cephalic configurations.
* Vein mapping studies completed 2.5-3 mm minimum vein diameter on mapping.

Exclusion Criteria:

* Ipsilateral proximal venous and arterial occlusion or stenosis
* systemic or local infection at the site planned for AVF creation.
* Anticipated inability to keep 30-day post-operative follow-up appointment.
* Revision AVF, Synthetic graft AVF, or lower limb AVF.
* Patients with absent distal pulses and chronic ischemia of the upper limb.
* Recent cannulation of puncture of the vein within two weeks before its use in AVF creation.
* Vasculitis (collagen diseases)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Functional Maturation of Arterio-venous Fistula | 6 months
  The suitability of an AVF for successful cannulation for dialysis, ascertained by duplex ultrasound study by measuring vein length at least 10 cm, diameter more than 6 mm, depth for skin not more than 6 mm, and ability of the access to deliver a flow rate of 600ml/min and maintain dialysis for 4 hours.

SECONDARY OUTCOMES:
Complication rate and failure of maturation | Six Months
  Bleeding, infection, steal syndrome, and aneurysmal dilatation at the anastomosis site.

CONTACTS AND LOCATIONS:
Overall Officials: ahmed fouda, MD, Principal Investigator — Kafrelsheikh University
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Coresh J, Selvin E, Stevens LA, Manzi J, Kusek JW, Eggers P, Van Lente F, Levey AS. Prevalence of chronic kidney disease in the United States. JAMA. 2007 Nov 7;298(17):2038-47. doi: 10.1001/jama.298.17.2038. PMID 17986697
- [Background] Ibbotson SH, Walmsley D, Davies JA, Grant PJ. Generation of thrombin activity in relation to factor VIII:C concentrations and vascular complications in type 1 (insulin-dependent) diabetes mellitus. Diabetologia. 1992 Sep;35(9):863-7. doi: 10.1007/BF00399933. PMID 1397782
- [Background] Pozzoni P, Del Vecchio L, Pontoriero G, Di Filippo S, Locatelli F. Long-term outcome in hemodialysis: morbidity and mortality. J Nephrol. 2004 Nov-Dec;17 Suppl 8:S87-95. PMID 15599892
- [Background] Lee CP, Chertow GM, Zenios SA. An empiric estimate of the value of life: updating the renal dialysis cost-effectiveness standard. Value Health. 2009 Jan-Feb;12(1):80-7. doi: 10.1111/j.1524-4733.2008.00401.x. PMID 19911442
- [Background] Baboolal K, McEwan P, Sondhi S, Spiewanowski P, Wechowski J, Wilson K. The cost of renal dialysis in a UK setting--a multicentre study. Nephrol Dial Transplant. 2008 Jun;23(6):1982-9. doi: 10.1093/ndt/gfm870. Epub 2008 Jan 3. PMID 18174268
- [Background] Johansen KL, Chertow GM, Gilbertson DT, Herzog CA, Ishani A, Israni AK, Ku E, Li S, Li S, Liu J, Obrador GT, O'Hare AM, Peng Y, Powe NR, Roetker NS, St Peter WL, Saeed F, Snyder J, Solid C, Weinhandl ED, Winkelmayer WC, Wetmore JB. US Renal Data System 2021 Annual Data Report: Epidemiology of Kidney Disease in the United States. Am J Kidney Dis. 2022 Apr;79(4 Suppl 1):A8-A12. doi: 10.1053/j.ajkd.2022.02.001. No abstract available. PMID 35331382
- [Background] Lok CE, Huber TS, Lee T, Shenoy S, Yevzlin AS, Abreo K, Allon M, Asif A, Astor BC, Glickman MH, Graham J, Moist LM, Rajan DK, Roberts C, Vachharajani TJ, Valentini RP; National Kidney Foundation. KDOQI Clinical Practice Guideline for Vascular Access: 2019 Update. Am J Kidney Dis. 2020 Apr;75(4 Suppl 2):S1-S164. doi: 10.1053/j.ajkd.2019.12.001. Epub 2020 Mar 12. PMID 32778223
- [Background] Celik S, Gok Oguz E, Ulusal Okyay G, Selen T, Ayli MD. The impact of arteriovenous fistulas and tunneled cuffed venous catheters on morbidity and mortality in hemodialysis patients: A single center experience. Int J Artif Organs. 2021 Apr;44(4):229-236. doi: 10.1177/0391398820952808. Epub 2020 Sep 22. PMID 32962489
- [Background] Bray BD, Boyd J, Daly C, Donaldson K, Doyle A, Fox JG, Innes A, Khan I, Peel RK, Severn A, Shilliday I, Simpson K, Stewart GA, Traynor J, Metcalfe W; Scottish Renal Registry. Vascular access type and risk of mortality in a national prospective cohort of haemodialysis patients. QJM. 2012 Nov;105(11):1097-103. doi: 10.1093/qjmed/hcs143. Epub 2012 Aug 20. PMID 22908320
- [Background] Lin PH, Bush RL, Nguyen L, Guerrero MA, Chen C, Lumsden AB. Anastomotic strategies to improve hemodialysis access patency--a review. Vasc Endovascular Surg. 2005 Mar-Apr;39(2):135-42. doi: 10.1177/153857440503900202. PMID 15806274
- [Background] Achneck HE, Sileshi B, Li M, Partington EJ, Peterson DA, Lawson JH. Surgical aspects and biological considerations of arteriovenous fistula placement. Semin Dial. 2010 Jan-Feb;23(1):25-33. doi: 10.1111/j.1525-139X.2009.00651.x. PMID 20331815
- [Background] Konner K, Lomonte C, Basile C. Placing a primary arteriovenous fistula that works--more or less known aspects, new ideas. Nephrol Dial Transplant. 2013 Apr;28(4):781-4. doi: 10.1093/ndt/gfs463. Epub 2012 Nov 2. PMID 23125423